CLINICAL TRIAL: NCT05459376
Title: Effect of Dry Cupping Therapy Associated With the McKenzie Method in Patients With Chronic Low Back Pain: Protocol for a Sham-controlled Randomized Trial
Brief Title: Effect of Dry Cupping Therapy Associated With the McKenzie Method in Patients With Chronic Low Back Pain
Acronym: MDTDryCup
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Adjunct Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRNMDTDryCupping
Record Dates: First submitted 2022-07-11; First posted 2022-07-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention Group and Sham Group
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessments will be carried out by researcher A who will not be involved with the interventions and will remain blind to the identification of groups.
  Each participant will remain identified by numbers and not names. Participants will be informed about the aim of the study to assess the additional effect of two different cupping techniques, the classic and the sham, in association with active exercise. In order not to compromise the blinding of the study, all participants will undergo the same assessment before the interventions. Intervention times will be differentiated so that there is no contact between the groups and possible exchanges of information. Data collected during participant assessments will not be revealed to the researchers responsible for the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive an assessment, classification as to McKenzie method (MDT) syndrome and indication of the preferred direction of movement, whether flexion, extension or lateral displacement of the spine ; will receive basic information about low back pain (LBP), its prevalence and prognosis; plus how and why to exercise; and types of responses that may occur in response to the exercise program. Guidance for performing the exercises at home. Dry suction cup application with 6 size 1 acrylic cups (4.5 cm internal diameter) with a distance of 3 cm each cup, parallel to the L1 to L5 vertebrae, bilaterally according to the acupoint boundaries, B23, B24 and B25 . This group will consist of performing MDT exercises and dry cupping with 2 suctions for 10 minutes, 2 times a week, for 8 weeks.
  Interventions: Other: Exercises and dry cupping
- Sham Group (Sham Comparator): The sham group will follow the same principles of evaluation, classification and intervention according to the McKenzie method (MDT) (described in the intervention group) and will have a placebo dry cup application with 6 size 1 acrylic cups (4.5 cm internal diameter) with a distance of 3 cm each cup, parallel to the vertebrae L1 to L5, bilaterally . This group will consist of placebo dry cupping for 10 minutes, 2 times a week, for 8 weeks. However, cups will be prepared with small holes <2 mm in diameter to release negative pressure in seconds.
  Interventions: Other: Exercises and dry cupping

INTERVENTIONS:
Other: Exercises and dry cupping — Participants in the intervention group will receive an assessment, classification as to MDT syndrome and indication of the preferred direction of movement, whether flexion, extension or lateral displacement of the spine
  Other Names: exercises

SUMMARY:
Introduction: Currently, clinical practice guidelines recommend exercise as a first-line approach to the treatment of chronic low back pain (LBP). On the other hand, passive techniques such as cupping therapy have gained space in the management of this population, however, important gaps regarding the combination of cupping therapy with active exercises in individuals with nonspecific chronic low back pain are still present in the literature. In this context, this protocol describes a sham-controlled, randomized and blinded study that aims to evaluate the additional effects of cupping therapy in association with McKenzie method exercises on pain and functional outcomes of individuals with nonspecific chronic low back pain. Methods: 108 individuals with nonspecific and localized chronic low back pain in the age group of 18 to 59 years will be recruited and evaluated, regarding the inclusion and exclusion criteria. Subsequently, they will be randomized to one of 2 groups: intervention group, in which they will be submitted to the McKenzie method intervention and later the addition of the dry suction cup; and sham group, in which, after the intervention of the McKenzie method, the application of the sham cup will be added.

DETAILED DESCRIPTION:
The individuals will be classified and treated according to the McKenzie method (MDT) and then they will receive the application of cups in parallel to the vertebrae from L1 to L5, bilaterally. Interventions will be carried out twice a week for eight weeks. Volunteers will be evaluated before treatment (T0), immediately after the first intervention (T1), with 4 weeks of intervention (T4) and with 8 weeks of intervention (T8)

The individuals will be classified and treated according to the McKenzie method and then they will receive the application of cups in parallel to the vertebrae from L1 to L5, bilaterally. Interventions will be carried out twice a week for eight weeks. Volunteers will be evaluated before treatment (T0), immediately after the first intervention (T1), with 4 weeks of intervention (T4) and with 8 weeks of intervention (T8). The primary outcome will be physical function, functionality (Timed Up and Go test), while the secondary outcomes will be pain intensity (Numerical Pain Scale), lumbar range of motion (finger to floor test), patient expectation and patient perception (Global Perceived Effect Scale).

ELIGIBILITY:
Inclusion Criteria:

* Individuals, male and female, 18 to 59 years, non-obese, with non-specific localized LBP for more than 3 months;
* Report pain intensity between 3 and 8 according to the numerical pain scale;

Exclusion Criteria:

* Have previously performed cupping therapy in some body segment;
* Present neurological, vestibular, visual or auditory deficits that make assessments impossible;
* Being in the gestational period;
* Having severe spinal disease (including fractures, tumour, inflammatory diseases, or tumours);
* Have undergone previous spinal surgery;
* Present with radiating or sacroiliac back pain; another rheumatic disease such as fibromyalgia,or ankylosing spondylitis.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Disability - ODI | baseline and 8 weeks after
  The Oswestry Disability Index (ODI) questionnaire will be used to analyze disability in people with low back pain.This instrument contains 10 items that assess the impact of low back pain on various functional activities. Values range from 0 to 5, with the highest value indicating greater disability. The final result is the sum of all items. The validated version in Portuguese is used.

SECONDARY OUTCOMES:
Change Numerical Pain Scale - NPS | baseline, immediately after 1 intervention, 4 and 8 weeks after the intervention
  The pain will be measured by the Numerical Pain Scale (NPS). Patients will be asked to circle the number between 0 and 10, zero represents "no pain", while the upper limit represents "the worst possible pain". The NPS score will be collected with the individual at rest, during the assessment of trunk range of motion and during the execution of the Timed Up and Go test.
Change in Functional test - Timed Up and Go (TUG) | baseline and 8 weeks after
  Functional test: Timed Up and Go (TUG): is a functional test that quantifies the mobility of an individual in seconds through the time he performs the task, that is, how many seconds he gets up from a chair, walks 3 meters, turns, goes back to the chair and stands again. The test was primarily designed to assess risk of falls in the elderly, with the following scores: less than 20 seconds for performance, corresponding to low risk of falling, 20 to 29 seconds, medium risk of falls, and 30 seconds or more, a high risk of falling. The subject will take the test 3 times and the average of the 3 trials will be noted.
Change in Trunk range of motion - Range of motion (ROM) | baseline, immediately after 1 intervention, 4 and 8 weeks after the intervention
  Trunk range of motion: Range of motion (ROM) will be measured using the finger-to-floor test. It has high reliability and can be used for clinical practice and scientific studies.The finger-to-floor test is performed with the subject standing upright and with feet together. The participant will be asked to lean forward as much as possible, keeping the knees, arms and fingers fully extended. The vertical distance between the tip of the middle finger and the floor is measured with a tape measure.
Change in participant perception | baseline and 8 weeks after
  The Brazilian version of the Global Perceived Effect Scale will assess participant self-perception of interventions. It uses a scale of 11 points ranging from a negative five (extremely worse) to a positive five (completely recovered) compared with baseline
Change in participant expectation | baseline
  A Likert-type scale will be used to assess the expectation of participants regarding the treatment. The following question will be used: "Do you think that with the application of dry cupping therapy, you will: (1) get much worse, (2) get a little worse, (3) get neithe better nor worse, (4) get a little better, or (5) get a lot better."

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C de Souza, PT, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Marcelo Cardoso de Souza, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Almeida Silva HJ, Barbosa GM, Scattone Silva R, Saragiotto BT, Oliveira JMP, Pinheiro YT, Lins CAA, de Souza MC. Dry cupping therapy is not superior to sham cupping to improve clinical outcomes in people with non-specific chronic low back pain: a randomised trial. J Physiother. 2021 Apr;67(2):132-139. doi: 10.1016/j.jphys.2021.02.013. Epub 2021 Mar 20. PMID 33757719
- [Background] Almeida Silva HJ, Avila MA, Castro KMS, Pinheiro YT, Lins CAA, Medeiros Barbosa G, de Souza MC. Exploring patient experiences of participating in a real and sham dry cupping intervention for nonspecific low back pain: A qualitative study. PLoS One. 2022 May 19;17(5):e0268656. doi: 10.1371/journal.pone.0268656. eCollection 2022. PMID 35587506
- [Derived] da Silva KMP, Almeida Silva HJ, Pontes-Silva A, DeSantana JM, Avila MA, Barbosa GM, de Souza MC. What are the effects of dry cupping therapy combined with the McKenzie method on clinical outcomes in chronic low back pain? A protocol for a randomized, sham-controlled trial. BMC Complement Med Ther. 2025 Jul 2;25(1):219. doi: 10.1186/s12906-025-04940-9. PMID 40604805